CLINICAL TRIAL: NCT02201485
Title: Balloon Angioplasty Alone Versus in Combination With Stent Placement for the Treatment of Budd-Chiari Syndrome in China: An Randomized Controlled Trial
Brief Title: Budd-Chiari Syndrome in China: Balloon Angioplasty Alone or Combined With Stent Placement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2BCS-rencanalization
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Budd-Chiari Syndrome
Keywords: Budd-Chiari syndrome; percutaneous recanalization; treatment; reocclusion; patency
MeSH Terms: conditions — Budd-Chiari Syndrome | interventions — Stents

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTA in combination with stent-placement (Active Comparator): In this group, the patients will undergo percutaneous balloon angioplasty with or without stent-placement angioplasty in combination with stent-placement.
  Interventions: Device: Stent; Device: Balloon
- PTA alone (Active Comparator): In this group, the patients will undergo percutaneous balloon angioplasty alone. The patients will transfer to the stent placement in the following cases: 1) reocclusion with thrombosis; and 2) at least 2 reocclusion events.
  Interventions: Device: Balloon

INTERVENTIONS:
Device: Stent
  Arms: PTA in combination with stent-placement
Device: Balloon

SUMMARY:
Budd-Chiari syndrome (BCS) is defined as the hepatic outflow obstruction from the small hepatic veins to the confluence between inferior vena cava and right atrium, which often leads to the life-threatening complications, such as liver failure and portal hypertension-related complications. At present, a stepwise treatment strategy is employed, including anticoagulation, thrombolysis, percutaneous recanalization (i.e., percutaneous transluminal angioplasty [PTA] alone or in combination with stent placement), transjugular intrahepatic portosystemic shunt, and liver transplantation. In West, only less than 20% of BCS patients underwent percutaneous recanalization; by contrast, percutaneous recanalization is the most common treatment modality used in China.

Recently, an 11-year retrospective case series of 177 Chinese patients with primary BCS has shown a higher rate of re-occlusion in the PTA alone group than in the PTA combined with stent placement group (31% versus 7.7%, p<0.001). In addition, re-occlusion was regarded as the independent predictor of mortality. Accordingly, we hypothesized that PTA alone might have a worse survival than PTA combined with stent placement in Chinese patients with primary BCS.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age 18-75 years old.
3. Budd-Chiari syndrome
4. Child-Pugh score <13 points.
5. Eligible for percutaneous recanalization.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Malignancy.
3. HIV infection.
4. Severe cardiac or lung diseases.
5. Severe renal dysfunction (serum> 265.2 umol/l).
6. Uncontrolled systemic infection.
7. Allergic to contrast agents.
8. Poor compliance.
9. A prior history of percutaneous recanalization.
10. Ineligible for percutaneous recanalization.
11. Liver cirrhosis with severe portal hypertension-related complications.
12. Acute liver failure.
13. Progressive deterioration of liver function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-05; Primary Completion 2017-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
The incidence of reocclusion between PTA alone and in combination with stent-placement groups | 2 years

SECONDARY OUTCOMES:
The survival between PTA alone and in combination with stent placement groups | 2 years
The incidence of procedure-related complications between PTA alone and in combination with stent placement groups | 2 years
The length of hospitalization between PTA alone and in combination with stent placement groups | 2 years
The symptom recurrence rate between PTA alone and in combination with stent placement groups | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi’an, Shanxi, China

REFERENCES:
- [Background] Han G, Qi X, Zhang W, He C, Yin Z, Wang J, Xia J, Xu K, Guo W, Niu J, Wu K, Fan D. Percutaneous recanalization for Budd-Chiari syndrome: an 11-year retrospective study on patency and survival in 177 Chinese patients from a single center. Radiology. 2013 Feb;266(2):657-67. doi: 10.1148/radiol.12120856. Epub 2012 Nov 9. PMID 23143028
- [Background] Qi X, Han G. Images in clinical medicine. Abdominal-wall varices in the Budd-Chiari syndrome. N Engl J Med. 2014 May 8;370(19):1829. doi: 10.1056/NEJMicm1308567. No abstract available. PMID 24806162
- [Background] Qi X, Wu F, Ren W, He C, Yin Z, Niu J, Bai M, Yang Z, Wu K, Fan D, Han G. Thrombotic risk factors in Chinese Budd-Chiari syndrome patients. An observational study with a systematic review of the literature. Thromb Haemost. 2013 May;109(5):878-84. doi: 10.1160/TH12-10-0784. Epub 2013 Feb 28. PMID 23447059
- [Background] Qi X, Wu F, Fan D, Han G. Prevalence of thrombotic risk factors in Chinese Budd-Chiari syndrome patients: results of a prospective validation study. Eur J Gastroenterol Hepatol. 2014 May;26(5):576-7. doi: 10.1097/MEG.0000000000000056. No abstract available. PMID 24694738
- [Background] Qi X, Guo W, He C, Zhang W, Wu F, Yin Z, Bai M, Niu J, Yang Z, Fan D, Han G. Transjugular intrahepatic portosystemic shunt for Budd-Chiari syndrome: techniques, indications and results on 51 Chinese patients from a single centre. Liver Int. 2014 Sep;34(8):1164-75. doi: 10.1111/liv.12355. Epub 2013 Nov 20. PMID 24256572
- [Background] Qi X, Han G, Guo W, Yin Z, Fan D. Education and Imaging. Hepatobiliary and pancreatic: Budd-Chiari syndrome with infra-hepatic obstruction of inferior vena cava. J Gastroenterol Hepatol. 2013 Jun;28(6):905. doi: 10.1111/jgh.12228. No abstract available. PMID 23692579
- [Derived] Wang Q, Li K, He C, Yuan X, Luo B, Qi X, Guo W, Bai W, Yu T, Fan J, Wang Z, Yuan J, Li X, Zhu Y, Han N, Niu J, Lv Y, Liu L, Li J, Tang S, Guo S, Wang E, Xia D, Wang Z, Cai H, Wang J, Yin Z, Xia J, Fan D, Han G. Angioplasty with versus without routine stent placement for Budd-Chiari syndrome: a randomised controlled trial. Lancet Gastroenterol Hepatol. 2019 Sep;4(9):686-697. doi: 10.1016/S2468-1253(19)30177-3. Epub 2019 Jul 3. PMID 31279647